CLINICAL TRIAL: NCT03380052
Title: The Evaluation of OLGA and OLGIM Stage Systems for Prediction of Gastric Cancer Risk and Interaction With Other Risk Factors According to Lauren's Classification
Brief Title: OLGA and OLGIM Stage System for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1610/368-106
Record Dates: First submitted 2017-12-16; First posted 2017-12-20 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stomach Neoplasms; Atrophic Gastritis; Intestinal Metaplasia
Keywords: OLGA; OLGIM; Helicobacter pylori; Gastric cancer; pepsinogen
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer: Patients who were diagnosed with gastric cancer
- Control: Healthy participants or benign disease patients such as benign gastric ulcers, duodenal ulcers, reflux esophagitis, or non-erosive reflux disease

SUMMARY:
To validate OLGA and OLGIM staging system with serum pepsinogen for estimating GC risk according to Lauren's histologic classification in South Korea. Also attempted to estimate synergistic interaction among the several risk factors to help establish surveillance strategy.

DETAILED DESCRIPTION:
To validated the OLGA and OLGIM staging system with serum pepsinogen to estimate gastric cancer risk according to Lauren's histologic classification in South Korea, where the incidence rate of GC is high. In addition, the investigators attempted to investigate the interaction among the several risk factors including OLGA or OLGIM staging system for the risk of GC to help establish surveillance strategy.

ELIGIBILITY:
Inclusion Criteria:

* Control group

  * those who were between 25 and 80 years old and did not have any evidence of gastric cancer and gastric dysplasia, esophageal tumor and MALToma in upper gastrointestinal endoscopy
* Gastric cancer group

  * Patients diagnosed as gastric cancer in the upper gastrointestinal endoscopy at the time of participating in the study between 25 and 80 years old.

Exclusion Criteria:

* history of previous gastrointestinal surgery,
* any other malignancy
* cardia cancer
* who do not perform endoscopic biopsy
* pathologically proven gastric dysplasia

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visited gastroenterology department complaining of gastrointestinal symptoms and underwent esophagogastroduodenoscopy (EGD)
Sampling Method: Probability Sample
Enrollment: 2900 (Actual)
Dates: Start 2006-02 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of OLGA and OLGIM stage systems with serum pepsinogen for prediction of gastric cancer risk | per 1 year
  To validate OLGA and OLGIM staging system with serum pepsinogen for estimating GC risk according to Lauren's histologic classification

CONTACTS AND LOCATIONS:
Overall Officials: Officials Officials, Officials, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No